CLINICAL TRIAL: NCT04801043
Title: A Phase 1, Single-Dose, Randomized, Double Blind, Placebo-Controlled Study to Evaluate Pharmacokinetics, Safety and Tolerability of XNW4107 for Injection in Healthy Adult Young Females and in Healthy Adult Elderly Males and Females.
Brief Title: To Evaluate the Pharmacokinetics of XNW4107 in Healthy Adult Young Females and in Healthy Adult Elderly Males and Females.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Evopoint Biosciences Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: XNW4107-002
Record Dates: First submitted 2021-03-07; First posted 2021-03-16 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Bacterial Infections
MeSH Terms: conditions — Bacterial Infections | interventions — Cilastatin, Imipenem Drug Combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1: Healthy young females (Experimental): Healthy young females participants, ≥ 18 to ≤ 45 years of age, randomized to receive a single dose of XNW4107 250mg IV co-administered with imipenem 500mg /cilastatin 500mg.
  Interventions: Drug: XNW4107; Drug: Imipenem/Cilastatin
- Cohort 2: Healthy elderly males (Experimental): Healthy elderly male participants, ≥ 65 years of age, randomized to receive a single dose of XNW4107 250mg IV co-administered with imipenem 500mg /cilastatin 500mg.
  Interventions: Drug: XNW4107; Drug: Imipenem/Cilastatin
- Cohort 3: Healthy elderly females (Experimental): Healthy elderly female participants, ≥ 65 years of age, randomized to receive a single dose of XNW4107 250mg IV co-administered with imipenem 500mg /cilastatin 500mg.
  Interventions: Drug: XNW4107; Drug: Imipenem/Cilastatin
- Placebo to XNW 4107 & imipenem/cilastatin (Placebo Comparator): Matching placebo for XNW4107 and imipenem/cilastatin
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: XNW4107 — XNW4107 250mg IV over 60 minutes as a single dose
  Arms: Cohort 1: Healthy young females; Cohort 2: Healthy elderly males; Cohort 3: Healthy elderly females
Drug: Imipenem/Cilastatin — 500mg/500mg IV over 60 minutes as a single dose
  Arms: Cohort 1: Healthy young females; Cohort 2: Healthy elderly males; Cohort 3: Healthy elderly females
Drug: placebo — Matching placebo to XNW4107 containing the same inactive ingredients IV over 60 minutes as a single dose
  Matching placebo to Imipenem/Cilastatin 0.9% sodium chloride IV over 60 minutes as a single dose
  Arms: Placebo to XNW 4107 & imipenem/cilastatin

SUMMARY:
This is a Phase 1, randomized, double-blind, placebo-controlled study to assess the PK, safety and tolerability of XNW4107, imipenem and cilastatin administered by 60-min (± 3 min) IV infusion in healthy adult young females and in healthy adult elderly males and females.

ELIGIBILITY:
Inclusion Criteria:

* 1. Healthy adult female, 18 to 45 years of age (both inclusive) or 65 years or over (≥ 65 years); or healthy adult male 65 years or over (≥ 65 years).

  2. BMI ≥ 18.0 and ≤ 32.0 (kg/m²) and weight between 55.0 and 100.0 kg (inclusive).

  3. Medically healthy without clinically significant abnormalities as assessed by the Investigator based on Screening medical history, physical examination, vital signs, 12-lead ECG, hematology, biochemistry and urinalysis.

  4. Male or female, willing to contracept. If female, must be non-pregnant and non-lactating.

  5. Ability and willingness to abstain from alcohol, caffeine, xanthine-containing beverages or food (coffee, tea, chocolate, and caffeine-containing sodas, colas, etc.) or product containing any of these from 48 hours prior to study drug administration until discharge from the clinical unit.

Exclusion Criteria:

* 1. History or presence of significant oncologic, cardiovascular, pulmonary, hepatic, renal, hematological, gastrointestinal, endocrine, immunologic, dermatologic, vascular or neurological disease, including any acute illness or surgery within the past 3 months determined by the Investigator to be clinically relevant.

  2. Electrocardiogram (ECG) with QTcF interval duration equal or greater than 450 msec for males and 470 msec for females obtained after at least 5 minutes in a supine or semi-supine position at quiet rest at Screening or Check-In (Day -1).

  3. Subjects who have any of the following abnormalities on laboratory values at Screening or prior confinement including: • White blood cell count < 3,000/mm³, hemoglobin < 11g/dL; • Absolute neutrophil count <1,200/mm³, platelet count <120,000/mm³; • Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) greater than 1.5 x the upper limit of normal (ULN) for the reference laboratory.

  4. History of seizure disorder except childhood history of febrile seizures.

  5. Positive testing for severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) at Screening.

  6. Close contact with anyone who tested positive for SARS-CoV-2 infection, or presence of symptoms associated with SARS-CoV-2 infection at Screening or Check-in, or within 14 days prior to Screening.

  7. Recent history (within 6 months) of known or suspected Clostridium difficile infection.

  8. Positive testing for HIV Ab, HBsAg or HCV Ab.

  9.Positive urine drug or alcohol testing at screening or check-in (Day -1).

  10.Use of prescription medications (with the exception of hormone replacement therapy and contraceptives), including nonsteroidal anti-inflammatory drugs, sucralfate, or herbal preparations within 7 days before Check in (Day -1), or use of an over-the-counter medication, acetaminophen (>2 g/day), vitamins, or supplements (including fish liver oils) within 7 days before Check in (Day -1); or probenecid or valproic acid within 30 days before Check in (Day -1).

  11. Receipt of an investigational drug within 30 days or 5 half-lives prior to the first administration of study drug, whichever is longer.

  12. Known history of clinically significant hypersensitivity reaction or anaphylaxis to any medication, or history of clinically significant hypersensitivity to the study drug or any related drugs or to any of the excipients, or significant food intolerance.

  13. Donation of blood or plasma within 30 days prior to dosing, or loss of whole blood of more than 500 mL within 30 days prior to dosing, or receipt of a blood transfusion within 1 year of study enrollment.

  14. Any other condition or prior therapy, which, in the opinion of the Investigator, would make the volunteer unsuitable for this study, including inability to cooperate fully with the requirements of the study protocol or likely to be non-compliant with any study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-03-02 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
(Plasma)Total body clearance (CL/F) of of XNW4107, imipenem and cilastatin. | From baseline to 48 hours post-dose
(Plasma) Area under the curve from time zero to the last quantifiable sample (AUC0-last) of XNW4107, imipenem and cilastatin. | From baseline to 48 hours post-dose
(Plasma) AUC extrapolated to infinity (AUC0-∞) of of XNW4107, imipenem and cilastatin. | From baseline to 48 hours post-dose
(Plasma) Apparent steady-state volume of distribution (Vss/F) of of XNW4107, imipenem and cilastatin. | From baseline to 48 hours post-dose
(Plasma) Maximum plasma concentration (Cmax) of of XNW4107, imipenem and cilastatin. | From baseline to 48 hours post-dose
(Plasma) Time to the maximum plasma concentration (Tmax) of of XNW4107, imipenem and cilastatin. | From baseline to 48 hours post-dose
(Plasma) The terminal elimination half-life (t1/2) of XNW4107, imipenem and cilastatin. | From baseline to 48 hours post-dose
(Urine) Renal clearance (CLR) of the XNW4107, imipenem and cilastatin dose administered. | From baseline to 48 hours post-dose
(Urine) Fraction of drug excreted in the urine expressed as a percentage of the XNW4107, imipenem and cilastatin dose administered (Ae%) | From baseline to 48 hours post-dose
(Urine) Amount of drug excreted in the urine through 24 hours (Ae0-24) | From baseline to 24 hours post-dose
(Urine) Amount of drug excreted in the urine through 48 hours (Ae0-48) | From baseline to 48 hours post-dose

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events of Hematology as assessed by CTCAE v5.0 | From baseline up to 10 days post-dose
  Safety and tolerability up to the last study visit as assessed by the incidence of treatment-emergent AEs along with clinically significant changes from baseline in clinical laboratory values of Hematology including White cell count with differential (total and % of neutrophil, lymphocyte, monocyte, eosinophil, and basophil), red blood cell count in m/mm³, hemoglobin in g/dL, hematocrit in %, mean corpuscular volume and platelet count m/mm³.
Number of participants with treatment-related adverse events of Physical Examination as assessed by CTCAE v5.0. | From baseline up to 10 days post-dose
  Safety and tolerability up to the last study visit as assessed by the incidence of treatment-emergent AEs along with clinically significant changes from baseline in Physical Examination of the following body systems: HEENT; cardiovascular, respiratory, gastrointestinal, dermatological, musculoskeletal, nervous systems, lymph nodes and general appearance, and in kilograms, height in meters and weight and height will be combined to report BMI in kg/m².
Number of participants with treatment-related adverse events of Vital Signs as assessed by CTCAE v5.0. | From baseline up to 10 days post-dose
  Safety and tolerability up to the last study visit as assessed by the incidence of treatment-emergent AEs along with clinically significant changes from baseline in Vital Signs (Systolic and diastolic blood pressure in mmHg, heart rate in Beats per min, respiratory rate in Breaths per min, and oral temperature in Degree celsius).
Number of participants with treatment-related adverse events of 12-Lead Electrocardiogram (ECG) as assessed by CTCAE v5.0. | From baseline up to 3 days post-dose
  Safety and tolerability up to the last study visit as assessed by the incidence of treatment-emergent AEs along with clinically significant changes from baseline in 12-Lead Electrocardiogram including heart rate(bpm), RR interval(ms), PR interval(ms), QRS(ms), QT(ms) and QTcF(ms).
Number of participants with treatment-related adverse events of Biochemistry as assessed by CTCAE v5.0. | From baseline up to 10 days post-dose
  Safety and tolerability up to the last study visit as assessed by the incidence of treatment-emergent AEs along with clinically significant changes from baseline in clinical laboratory values of Biochemistry including Sodium in mmol/L, calcium in mg/dL, phosphate in mg/dL, potassium in mmol/L, chloride in mmol/L, glucose in mg/dl, BUN in mg/dl, uric acid in mg/dl, creatinine in mg/dL, creatine kinase in IU/L, creatinine clearance calculated in ml/min/1.73m² , total bilirubin in mg/dL, direct bilirubin in mg/dL, alkaline phosphatase in IU/L, ALT in IU/L, AST in IU/L, lactate dehydrogenase in IU/L, gamma-glutamyl transferase in IU/L, total protein in g/dL, albumin in g/dL, triglycerides in mg/dL, and cholesterol in mg/dL.
Number of participants with treatment-related adverse events of Coagulation as assessed by CTCAE v5.0. | From baseline up to 10 days post-dose
  Safety and tolerability up to the last study visit as assessed by the incidence of treatment-emergent AEs along with clinically significant changes from baseline in clinical laboratory values of Coagulation including Prothrombin time in seconds, activated partial thromboplastin time in seconds and International Normalized Ratio (INR).
Number of participants with treatment-related adverse events of Urinalysis as assessed by CTCAE v5.0. | From baseline up to 10 days post-dose
  Safety and tolerability up to the last study visit as assessed by the incidence of treatment-emergent AEs along with clinically significant changes from baseline in clinical laboratory values of Urinalysis Specific gravity, pH, leukocyte esterase, protein, glucose, ketones, bilirubin, blood, nitrite, urobilinogen.

CONTACTS AND LOCATIONS:
Locations (1):
- Orlando Clinical Research Center (OCRC), Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No